CLINICAL TRIAL: NCT05695443
Title: Oral Health in Prison: a Randomized Controlled Study of the Effect of Motivational Interview on Improving Prisoners' Oral Health
Brief Title: Oral Health in Prison: a Study on Improving Prisoners' Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oral Health Center of Expertise Rogaland, Norway (Other)
Collaborators: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OralHlthRogaland
Record Dates: First submitted 2022-11-22; First posted 2023-01-25 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Oral Health; Prisoners
Keywords: Oral health; Prisoner; Motivational Interviewing; Oral hygiene
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Following the initial oral examination and questionnaire, prisoners are randomly assigned into either a treatment or control group, blocking at prison level. The randomization tool at www.randomizer.org is used. Prisoners in the treatment group receive an up to 30 Motivational Interviewing conversation, aiming at improving oral health and oral health-related behavior. The intervention is carried out by dental staff in prison. Prisoners in the control group do not receive the MI intervention.
Who Masked: Participant, Care Provider
Masking Description: Prisoners are not informed whether they are in the treatment or control group and are therefore blind to treatment status. Dental staff is blind to prisoners' treatment status at the first oral examination and questionnaire. The prisoner's treatment status is revealed just after this. Hence, dental staff collects data prior to knowing the prisoners' treatment status, and only learns this when they start the MI-based conversation. When prisoners are back at T1 and T2 for follow-up oral examinations and questionnaires, dental staff might still remember whether the prisoner was treated or not. To partially account for potential bias in the oral examination (assessment of plaque and mucosal inflammation), there are two independent assessments of this at T1 and T2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (Experimental): Prisoners in this group are subjected to a MI-based conversation lasting up to 30 minutes aiming at improving oral health and oral health related behavior
  Interventions: Behavioral: Motivational Interviewing
- Control group (No Intervention): Prisoners in this group do not receive the MI-based intervention

INTERVENTIONS:
Behavioral: Motivational Interviewing — This study investigates the effects of an intervention based on Motivational Interviewing (MI) on oral hygiene, oral cleaning routines, and attitudes towards own oral health. The first step is for the dental staff to ask open questions to the prisoner about their oral health or oral health behavior. The next step is to confirm to the prisoner what he or she is doing. The third step is called reflection. At this stage, dental staff tries to provide reflections on what the prisoner have said, for example by repeating what the prisoner have said or say the same using synonyms (simple reflection), by extracting the underlying opinion or feeling (complex reflection), or by illuminate both negative and positive sides of the situation (double sided reflection). The final step is to summarize the conversation. In addition, the intervention includes a change plan, in which the prisoner and dental staff agrees on specific behavior that the prisoner should follow based on the MI conversation.
  Arms: Motivational Interviewing

SUMMARY:
This study investigates the effects of an intervention based on Motivational Interviewing (MI) on oral hygiene, oral cleaning routines, and attitudes toward own oral health of prisoners in Norway. Motivational Interviewing is a collaborative, person-centered form of guiding to elicit and strengthen motivation for change. All prisoners in the study undergo an oral examination to establish a baseline of oral health and a comprehensive questionnaire to identify risk factors and their attitudes towards their oral health and oral treatment. Norwegian-speaking prisoners are then randomized into either a treatment or control group. In the treatment group, dental staff initiate a conversation with the prisoner based on techniques from MI. Both groups finally receive a toilet bag with basic equipment to regularly clean their teeth. After 4 weeks and 12 weeks, prisoners are invited back for another oral examination and a follow-up questionnaire, to measure changes in oral hygiene, oral cleaning routines, and attitude toward their oral health. At four weeks a screening of general learning difficulties using the validated screening tool The Hayes Ability Screening Index (HASI) will be conducted. If the intervention proves to be an effective tool in improving oral hygiene, oral cleaning routines, and/or attitude towards own oral health, it can serve as an alternative proactive approach to improve the oral health of a vulnerable group in society. If the improvements in oral hygiene and oral cleaning routines are long-lasting, this may in turn lead to a reduced need for oral treatment. An improved attitude towards own oral health may, together with other rehabilitation programs in prison, improve the prisoner's self-esteem and chances to successfully returning to society after having served their prison sentence.

DETAILED DESCRIPTION:
Study design and procedures:

The geographic region of this study is Rogaland County in the southwestern part of Norway. There are four prisons in Rogaland County, all of which are included in the study. Three prisons are categorized as high-security prisons, and one is categorized as a low-security prison. The main difference between high and low-security prisons is the level of security measures, as prisoners in low-security prisons are allowed to move more freely within the prison. The low-security prison is mainly used for less serious criminal offenses, with a sentence time of between six months and two years. Those convicted to less than six months can apply to serve the time with an ankle bracelet, whereas those convicted for more than two years start serving in a high-security prison. However, many high-security prisoners are transferred to low-security prisons to serve the final part of their sentence. Hence, the population across prisons is likely to vary due to the severity of the criminal offense they have committed, especially across high and low-security prisons. However, as those with the least serious criminal offenses serve time with an ankle bracelet, and those with more severe convictions often serve the final part of their sentence in a low-security prison, the populations may not be that different from each other.

Recruitment procedures:

Recruitment is done somewhat differently across prisons, and different for those already imprisoned at the time of the start of data collection and those arriving in the prison during the data collection period. For those already imprisoned at the start of data collection, they are either informed about the study by prison officers or dental staff. This process should originally be done exclusively by prison officers, but capacity constraints forced us to use our own staff in two of the prisons. The information given is the same across all prisons, based on an information letter, which is also distributed to the prisoners. They then give their preliminary consent to participate within a couple of days after being informed.

Those who arrive at the prison during the period of data collection are either informed about the study by prison officers or prison health workers during their first days in prison. Again, recruitment is done depending on the capacity of prison officers. In one prison, the dental staff was involved in the recruitment process. The information provided is the same as for those already imprisoned, and they receive the same information letter. Prisoners give their preliminary consent to participate within a couple of days.

Formal consent is given to dental staff at the very beginning of their first meeting.

Data collection:

Data collection started in November 2021 and is likely to continue until the end of June 2023. There is funding to collect data one day a week in all four of the prison in the project period. If it turns out that it is difficult to recruit enough prisoners in one of the prisons, resources can be reallocated to one of the other prisons.

The end date for data collection depends, in addition to uncertainty regarding whether additional funding is approved, on the extent that the ongoing pandemic will affect data collection. If stricter infection control measures are enforced, prisons are likely to quickly deny access to external partners. The new omicron variant of the corona virus has already forced delays in three out of four prisons. During a period in which it is not possible for dental health personnel to enter a prison, it will be necessary to do follow-up examinations at times deviating from the times described below. It is also likely that there will be higher attrition during such periods, as prisoners are released or moved to a prison outside Rogaland County before it is possible to do follow-up examinations. Such attrition is independent of treatment status.

During the data collection period, it is an aim to recruit around 500 subjects. The number of subjects that is possible to recruit depends on several factors. First, there need to be enough people serving their prison sentences during the data collection period. Prisons in Rogaland County have not been fully occupied in recent years. Second, the proportion of prisoners who choose to participate is uncertain. Third, the time spent on each prisoner depends on how effectively the prison staff can bring prisoners to the examination room and how effective the routines of the dental staff are. Fourth, it is difficult to estimate how many of the prisoners have sufficient Norwegian language to participate in the study.

Each prisoner is followed for 12 weeks in total (first meeting T0, after 4 weeks, T1, and after 12 weeks, T2), and prisoners will continuously be recruited in the data collection period. The intervention occurs only at T0, and only for those randomized to the treatment group. During the first few months, those who are already imprisoned will be recruited, and once all of them have been given the chance to participate, the recruitment of new prisoners will start.

Data collection and sources of data:

Data collection will be carried out by trained dental staff inside the prisons during the data collection period. Most data collected will be on the individual (prisoner) level. Moreover, basic information about each of the four prisons in our study will also be collected.

The source of data will be a combination of clinical information from the oral examination, answers from the questionnaire, and a few observations done by dental staff during the consultation.

Clinical data will include information on decayed, missing, and filled teeth (DMFT). This data will only be collected at T0, as it is not possible to observe any change in these parameters during the follow-up period. Moreover, clinical data on plaque and mucosal inflammation will be collected, using the MPS index. This is our main variable of interest. Plaque is affected by oral hygiene routines and the intake of drinks and food that can damage teeth. Thus any observed difference in changes in plaque between the treatment group and the control group may be interpreted as an effect of the intervention. The dental staff has undergone a calibration exercise of both DMFT and MPS.

The questionnaire is extensive. It starts with some background questions about demographic and socio-economic status, which are not likely to change during the follow-up period, and thus only asked at T0. Next, questions about their views on their own oral health will be asked. In particular, they will be asked about how they perceive the condition of their own oral health, whether they want to improve it, whether they regularly visit a dentist outside of prison, their cleaning routines, and their intake of food and drinks. Some of these questions are secondary variables of interest. In the case of an intervention effect, prisoners may have an adjusted view of their oral health, and they may change their oral cleaning routines and intake of food and drinks. They will also be asked standardized questionnaires about their oral-health quality of life (OHPI-14) and their self-reported anxiety and discomfort with dental treatment (MDAS). As these are unlikely to change during the follow-up period, they are only asked at T0.

Data on their general physical and mental health will also be collected. To measure mental health, the standardized questionnaire Mental Health Inventory 5 (MHI-5) will be used. The MHI-5 questionnaire at all three meeting points will be conducted, as it is expected reduced effects of the intervention if they are experiencing worsened mental health. This may be important when studying heterogeneous effects of the intervention. Lastly, data on their alcohol and drug use (outside of prison) will be collected, using the short versions of the alcohol use disorders identification test (AUDIT-4) and the drug use disorders identification test (DUDIT), collected only at T0.

Dental staff also take note of how many times the prisoner asks questions about their findings from the oral examination. If the intervention raises their awareness of oral health, it is likely that those in the intervention group ask more questions during the follow-up period. Hence, this is also a second variable of interest.

Questions about what criminal offenses the prisoner had committed, and similar questions which could affect how safe dental staff would perceive the situation will not be asked. If, for example, the prisoner said that he was a convicted sexual offender or murderer, this could challenge the feeling of safety for the dental staff. In the consent to participate, the prisoners have approved that such information can be collected from the Norwegian Correctional Service. However, it is not certain that such administrative data are accessible to the research group.

Intervention:

Following the first examination (T0), the prisoners are randomized into treatment- or control group. The intervention is an up to 30 minutes conversation with the prisoner about his or her oral health, based on Motivational Interviewing. The intervention is carried out by dental staff in prison. Prior to the start of data collection, dental staff has been trained by MI-certified specialists from the Regional Alcohol and Drug Competence Center in Rogaland County. The training consisted of three days of seminar with group work and discussions, a practice MI conversation that has been recorded, transcribed and graded by the MI center in Bergen, and direct feedback on this practice conversation. In addition, guidance from a MI specialist at the Center for Alcohol and Drug Research at Stavanger University Hospital were available at all time if required by the dental staff.

The MI conversation follows the methodology of MI closely. The first step is for the dental staff to ask open questions to the prisoner, for example, "what cleaning routines do you have for your teeth?" or "what benefits could you get from brushing your teeth twice a day?". The next step is to confirm to the prisoner what he or she is doing, for example, "you are really trying hard to take good care of your teeth" or "you have managed to have good cleaning routines multiple times in the past". The third step is called reflection. At this stage, the dental staff tries to provide reflections on what the prisoner has said, for example by repeating what the prisoner has said or saying the same using synonyms (simple reflection), by extracting the underlying opinion or feeling (complex reflection), or by illuminate both negative and positive sides of the situation (double sided reflection). The final step is to summarize the conversation. In addition, the intervention included a change plan, in which the prisoner and dental staff agree on specific behavior that the prisoner should follow based on the MI conversation.

ELIGIBILITY:
Inclusion criteria:

* Everyone serving time in one of the four prisons during the period of the study (November 2021 to June 2023)
* Sufficient Norwegian language

Exclusion criteria:

- Insufficient Norwegian language

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Changes from baseline Mucosal-plaque index (MPS) | Baseline- 4 weeks-12 weeks
  A four-point plaque score (PS) and a four-point mucosal score (MS). For the PS, score of 1 suggests no visible plaque, score of 2 suggests plaque is barely visible, score of 3 suggests a moderate amount of plaque, and score of 4 suggests large amount of plaque almost covering the whole surface of teeth. For the MS, score of 1 suggests normal mucosal, score of 2 suggests mild inflammation, score of 3 suggests medium inflammation, and score of 4 suggests strong inflammation. For both scores, if in doubt between 1 and 2, they are instructed to score 1. If in doubt between 3 and 4, they are instructed to score 4. The index is designed to evaluate oral health and oral hygiene in groups of individuals. This makes it a suitable index to be used when conditions are not optimal to assess the patient. In prison, dental staff have limited equipment and poor light compared to an ordinary dental clinic. Therefore, using an index designed to be used outside of clinics was important.

SECONDARY OUTCOMES:
Questionnaire responses | Baseline- 4 weeks-12 weeks
  1. How would you rate your own dental health? Scores are measured on a five-point Likert-type scale from "very poor" to "very good"
  2. Dental care products used (toothbrush, toothpaste, mouthwash, floss, toothpicks)
  3. Drinking something added flavor/sugar during the last 4 weeks?
  4. Eating sweet foods during the last 4 weeks?
  5. Eaten/drinking sugary drinks outside of the main meals during the last 4 weeks?
  6. Use of "Change plan"
     Scores on 2-6 are measured on a six-point Likert-type scale from "several times a day" to "never")
  7. How have you felt the last 4 weeks (very anxious, been so far down that nothing has been able to cheer you up, calm and harmonious, down and sad,happy?) Scores are measured on a six-point Likert-type scale (1=all the time, 2=almost all the time, 3=a lot of the time, 4=part of the time, 5=a little part of the time, 6=not at all)

OTHER OUTCOMES:
Questions asked by the prisoner | Baseline-4 weeks-12 weeks
  Dental staff take notes of how many times the prisoner asks questions about his teeth. If the intervention successfully increases the prisoner's interest in his own oral health, we could expect more question about his oral health.

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke H Bull, PhD, Study Director — Oral Health Centre of Expertise, Stavanger
Locations (1):
- Norwegian Correctional Service, Sandnes, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bryne E, Bergum KH, Gjedrem WG. Improving Oral Health in Prisons (PriOH): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Dec 11;13:e60817. doi: 10.2196/60817. PMID 39661440

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT05695443/Prot_SAP_000.pdf